CLINICAL TRIAL: NCT03220009
Title: A Randomized Phase II Trial of Adjuvant Nivolumab or Expectant Observation Following Neoadjuvant Ipilimumab Plus Nivolumab and Surgical Resection of High-Risk Localized, Locoregionally Advanced, or Recurrent Mucosal Melanoma
Brief Title: Nivolumab or Expectant Observation Following Ipilimumab, Nivolumab, and Surgery in Treating Patients With High Risk Localized, Locoregionally Advanced, or Recurrent Mucosal Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was never approved by CTEP neither was it ever activated
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01239; NCI-2017-01239 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A091603 (Other: Alliance for Clinical Trials in Oncology); A091603 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2017-07-17; First posted 2017-07-18 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Cervical Carcinoma; Esophageal Carcinoma; Mucosal Melanoma; Mucosal Melanoma of the Head and Neck; Oral Cavity Mucosal Melanoma; Recurrent Melanoma; Stage II Vulvar Cancer AJCC v7; Stage III Vulvar Cancer AJCC v7; Stage IIIA Vulvar Cancer AJCC v7; Stage IIIB Vulvar Cancer AJCC v7; Stage IIIC Vulvar Cancer AJCC v7; Stage IV Oral Cavity Cancer AJCC v6 and v7; Stage IV Vulvar Cancer AJCC v7; Stage IVA Oral Cavity Cancer AJCC v6 and v7; Stage IVB Oral Cavity Cancer AJCC v6 and v7; Stage IVC Oral Cavity Cancer AJCC v6 and v7; Vaginal Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Esophageal Neoplasms; Melanoma; Vulvar Neoplasms; Vaginal Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Watchful Waiting; Observation; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (nivolumab, ipilimumab, surgery, active surveillance) (Active Comparator): PART I: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1. Within 3-6 weeks after receiving nivolumab and ipilimumab, patients undergo surgery per standard of care. Within 84 days of last surgical resection, patients may also undergo adjuvant RT, if clinically appropriate.
  PART II: Patients undergo active surveillance for 1 year.
  Interventions: Procedure: Conventional Surgery; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Patient Observation; Radiation: Radiation Therapy
- Arm II (nivolumab, ipilimumab, surgery, nivolumab) (Experimental): PART I: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1. Within 3-6 weeks after receiving nivolumab and ipilimumab, patients undergo surgery per standard of care. Within 84 days of last surgical resection, patients may also undergo adjuvant RT, if clinically appropriate.
  PART II: Patients receive nivolumab IV over 30 minutes once every 2 weeks for 4 doses. Patients then continue to receive nivolumab IV over 30 minutes once every 4 weeks for up to 11 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Conventional Surgery; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Conventional Surgery — Undergo surgery
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Patient Observation — Undergo active surveillance
  Other Names: Active Surveillance; deferred therapy; expectant management; observation; Watchful Waiting
  Arms: Arm I (nivolumab, ipilimumab, surgery, active surveillance)
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; RADIATION; Radiotherapeutics; radiotherapy; RT; Therapy, Radiation

SUMMARY:
This randomized phase II trial studies how well nivolumab or expectant observation following ipilimumab, nivolumab, and surgery work in treating patients with high-risk mucosal melanoma that is restricted to the site of origin without evidence of spread, has spread to a local and regional area of the body, or has come back. Monoclonal antibodies, such as nivolumab and ipilimumab, may interfere with the ability of tumor cells to grow and spread. Sometimes the mucosal melanoma may not need more treatment until it progresses. In this case, observation may be sufficient. It is not known if nivolumab or expectant observation following ipilimumab, nivolumab, and surgery may be better in treating patients with mucosal melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Recurrence free survival (RFS) in patients with mucosal melanoma (MM) treated with neoadjuvant ipilimumab plus nivolumab and surgery followed by adjuvant nivolumab and expectant observation.

SECONDARY OBJECTIVES:

I. Pathologic complete response with neoadjuvant ipilimumab plus nivolumab. II. Distant recurrence-free survival (DRFS) with adjuvant nivolumab and expectant observation.

III. Overall survival (OS) with adjuvant nivolumab and expectant observation. IV. Safety/toxicity as measured by maximum grade adverse event in (a) the neoadjuvant setting, (b) the adjuvant nivolumab cohort after randomization, and (c) the observation cohort after randomization.

V. Rate of delayed primary surgery.

TERTIARY OBJECTIVES:

I. Demonstrate that baseline tumors harboring a higher neoepitope burden have superior median RFS than those who have a lower neoepitope burden in the arm receiving adjuvant nivolumab.

II. Demonstrate that tumors with higher CD8+ infiltration at the tumor invasive margin at surgical resection have superior median RFS than those with lower CD8+ infiltration.

III. Demonstrate that tumors harboring a "T cell inflamed" ribonucleic acid (RNA) expression signature at surgical resection following neoadjuvant nivolumab plus ipilimumab have a superior distant RFS than those harboring a "non-T cell inflamed" signature, both in the overall group and within those who receive adjuvant nivolumab.

IV. Identify recurrent genetic alterations at baseline that are associated with higher CD8+/PD1+ infiltration at baseline and following 1 dose of neoadjuvant nivolumab plus ipilimumab.

V. Tumor response rate will be estimated based on patients whose imaging are captured and submitted during the neo-adjuvant portion of the study (imaging is not required).

OUTLINE:

PART I: Patients receive nivolumab intravenously (IV) over 30 minutes and ipilimumab IV over 30 minutes on day 1. Within 3-6 weeks after receiving nivolumab and ipilimumab, patients undergo surgery per standard of care. Within 84 days of last surgical resection, patients may also undergo adjuvant radiation therapy (RT), if clinically appropriate.

PART II: Within 84 days of last surgical resection, patients are randomized to 1 of 2 arms.

ARM I: Patients undergo active surveillance for 1 year.

ARM II: Patients receive nivolumab IV over 30 minutes once every 2 weeks for 4 doses. Patients then continue to receive nivolumab IV over 30 minutes once every 4 weeks for up to 11 doses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 90 days for 2 years, every 180 days for 3 years or until disease progression, whichever is first, and every 6 months thereafter until a maximum of 5 years following registration.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 ELIGIBILITY CRITERIA
* Documentation of disease:

  * Histologic documentation: histologically proven mucosal melanoma by local pathology
  * Tumor tissue: tumor tissue from the primary site of disease must be available for PD-L1 testing (stratification factor)
* Disease status

  * Tumors must have NOT been completely resected, or must be locoregionally recurrent if previously resected; tumor must be deemed potentially resectable by local surgeon
  * MM arising from the head/neck, genitourinary, or gastrointestinal tract
  * Disease meets any 1 of 4 characteristics:

    * Regional lymph node (LN) involvement; OR
    * Multifocal/satellite primary disease; OR
    * Single localized, primary disease meeting one of the following site-specific requirements:

      * Head/neck - any primary lesion if sinonasal; pT4a or above for nasal or oral cavity
      * Anorectal - any primary lesion
      * Conjunctiva - any primary lesion T2 or T3 stage by American Joint Committee on Cancer (AJCC)
      * Vaginal/cervical - any primary
      * Vulvar (hair bearing surface, labia majora) - AJCC cutaneous stage IIB or higher
      * Esophageal - any primary
    * Locoregionally recurrent following prior resection
  * No evidence of metastatic disease at the time of registration
* No prior medical therapy (chemotherapy, immunotherapy, biologic or targeted therapy) or radiation therapy for MM, unless locoregionally recurrent; if recurrent, no prior medical or radiation therapy is allowed for the latest recurrence
* No history of the following:

  * Active known or suspected autoimmune disease
  * Human immunodeficiency virus (HIV) with CD4+ count < 300 or detectable viral load; patients with HIV, undetectable viral load, and CD4+ count >= 300 are eligible
  * Known active hepatitis B or C

    * Hepatitis B can be defined as:

      * Hepatitis B virus surface antigen (HBsAg) > 6 months
      * Serum hepatitis B virus (HBV) deoxyribonucleic acid (DNA) 20,000 IU/ml (105 copies/ml), lower values 2,000-20,000 IU/ml (104-105 copies/ml) are often seen in hepatitis B virus e antigen (HBeAg)-negative chronic hepatitis B
      * Persistent or intermittent elevation in alanine aminotransferase (ALT)/aspartate aminotransferase (AST) levels
      * Liver biopsy showing chronic hepatitis with moderate or severe necroinﬂammation
    * Hepatitis C can be defined as:

      * Hepatitis C antibody (AB) positive
      * Presence of hepatitis C virus (HCV) RNA
  * Known active pulmonary disease with hypoxia defined as oxygen saturation < 85% on room air
* Not pregnant and not nursing

  * For women of childbearing potential only, a negative pregnancy test done =< 14 days prior to registration is required
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine clearance >= 30 mL/min by Modified Diet in Renal Disease (MDRD) equation or Cockcroft-Gault
* Total bilirubin =< 1.5 x upper limit of normal (ULN)

  * Except in case of Gilbert disease
* AST/ALT =< 2.5 x upper limit of normal (ULN)
* Thyroid-stimulating hormone (TSH) within normal limits (WNL)

  * Supplementation is acceptable to achieve a TSH WNL; in patients with abnormal TSH if free T4 is normal and patient is clinically euthyroid, patient is eligible
* Concomitant medications

  * No systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days of registration (inhaled steroids for patients with underlying chronic pulmonary disease is acceptable as long as they meet other eligibility as listed above)
  * No other planned concurrent investigational agents or other tumor directed therapy (chemotherapy, radiation) while on study
* STEP 2 ELIGIBILITY CRITERIA
* Surgical resection of all gross disease

  * This assessment will be made by the local investigator based on review of the operative report, pathology results, and/or radiology reports; microscopically positive margins (e.g. R1 resection) are permitted
* Completion of PD-L1 testing

  * Patients will be stratified as PD-L1 >= 5% versus (vs) < 5% OR inevaluable; baseline tumor will be utilized; if this returns inevaluable, efforts should be made to utilize the resected specimen
* Randomization within 112 days of completion of surgical

  * The primary region must be included on cross-sectional imaging (e.g. sinus/neck if arising from sinonasal primary; pelvis if genitourinary); radiographic changes considered nonspecific or possibly due to surgery or radiation are not considered evidence of disease
* No significant immune-related adverse event due to the nivolumab plus ipilimumab dose received in the neoadjuvant setting, as follows:

  * Any grade myocarditis, including an asymptomatic troponin elevation felt to be related to nivolumab plus ipilimumab
  * Any grade neurologic complication (e.g. meningitis, encephalitis, neuropathy); study chair should be contacted if there is any question whether an adverse event (AE) was neurologic in nature
  * Grade 2 or higher pneumonitis
  * Grade 2 colitis
  * Grade 2 or higher anemia (due to drug; unrelated anemia is not exclusionary)
  * Thyroid/adrenal AEs regardless of grade that have stabilized or are clinically asymptomatic are eligible
  * Fatigue, regardless of grade, is not a contraindication to randomization
  * Grade 4 AST or ALT elevation
  * Asymptomatic elevated amylase and lipase, regardless of grade, are not contraindications to randomization
  * Grade 4 rash; grade 3 rash is not a contraindication to randomization; any oropharyngeal lesions or bullous skin lesions that are suggestive of toxic epidermal necrolysis or Stevens-Johnson syndrome are contraindications to randomization regardless of the grade of rash

    * If not specified above, other Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher AEs deemed possibly related to the nivolumab plus ipilimumab are exclusions to randomization; AEs that were attributable to surgery or adjuvant RT would not be contraindications to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) | From randomization to either adjuvant nivolumab or observation until evidence of disease recurrence, assessed up to 5 years
  RFS of patients receiving adjuvant nivolumab will be compared to patients undergoing observation. Kaplan- Meier curves will be constructed and median RFS times will be calculated for each arm.

SECONDARY OUTCOMES:
Distant recurrence-free survival (DRFS) | From randomization to either adjuvant nivolumab or observation until a distant recurrence is observed, assessed up to 5 years
  Will be evaluated using the Kaplan- Meier method. Median times to DRFS will be calculated for each arm and a cox proportional hazards model will be constructed to determine if there is a DRFS benefit for patients in the adjuvant Nivolumab arm (compared to observation).
Incidence of adverse events evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 5 years
  Maximum grade adverse events will be summarized in each of the following settings: during the neo-adjuvant phase of the trial (i.e. from registration until a patient is randomized to adjuvant nivolumab or observation), the adjuvant nivolumab arm after randomization, he observation arm after randomization.
Overall survival (OS) | From randomization to either adjuvant nivolumab or observation until death due to any cause; assessed up to 5 years
  Will be evaluated using the Kaplan- Meier method. Median OS times will be calculated for each arm and a cox proportional hazards model will be constructed to determine if there is a DRFS benefit for patients in the adjuvant Nivolumab arm (compared to observation).
Rate of delayed surgery | Up to 6 weeks after registration
  Reasons for delay will be summarized and the rate of delay will be calculated along with a 95% confidence interval using the properties of the binomial distribution.

OTHER OUTCOMES:
CD8+ infiltration | Up to 5 years
  CD8+ infiltration levels will be compared to RFS times using a cox proportional hazards model.
Neoepitope burden | Up to 5 years
  Neoepitope burden will be compared to RFS using a cox proportional hazards model.
Pathologic complete response prior to surgery, for patients with imaging available | Up to time of surgery, assessed up to 5 years
  The rate of pathologic complete response will be estimated using and a 95% confidence interval will be calculated using properties of the binomial distribution.
Recurrent genetic alterations | Up to 5 years
  Patients will be categorized by driver mutation, including BRAF, RAS family (NRAS/KRAS/HRAS), KIT, and/or NF1 alterations. The degree of CD8+ and/or PD-L1 infiltration will be compared across various categories of driver mutation using descriptive statistics. Pending further advances in genomic understanding of these tumors, alternate categories may be constructed.
T cell inflammation | Up to 5 years
  Patients will be categorized has having a "T dell inflamed" RNA expression signature versus a "non-T cell inflamed" signature. These groups will be compared to each other in terms of RFS times using a cox proportional hazards model. An additional model will be constructed with randomized arm included to determine if there is an interaction between signature and arm.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Shoushtari, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (1):
- Alliance for Clinical Trials in Oncology, Boston, Massachusetts, United States